CLINICAL TRIAL: NCT02681120
Title: Pilot Study of the Effect of Weight Loss on Breast Tissue and Blood Biomarkers in Women at Increased Risk for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Tarah J Ballinger, MD (Other)
Responsible Party: Sponsor-Investigator, Tarah J Ballinger, MD, Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: IUSCC-0556; 1511957605 (Other: Indiana University IRB)
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Breast Neoplasms; Obesity
Keywords: Biomarkers; Breast imaging
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk/BMI > 30: Women at elevated risk for breast cancer will have imaging (MRI and mammogram) pre-bariatric surgery and 1 year post-bariatric surgery, and blood and tissue collection (blood draw and biopsy) pre-bariatric surgery, 2 weeks post-bariatric surgery, and 1 year post-bariatric surgery.
  Interventions: Procedure: Biopsy; Procedure: Blood draw; Procedure: Mammogram; Procedure: MRI
- Women with normal BMI: Deidentified samples that were donated to the IU Komen Tissue Bank will be used for comparison to the high risk/BMI > 30 cohort.

INTERVENTIONS:
Procedure: Biopsy
  Groups: High risk/BMI > 30
Procedure: Blood draw
  Groups: High risk/BMI > 30
Procedure: Mammogram
  Groups: High risk/BMI > 30
Procedure: MRI
  Groups: High risk/BMI > 30

SUMMARY:
This is a pilot, non-randomized, single institution, observational study investigating the effect of dramatic weight loss secondary to bariatric surgery on biomarkers of breast cancer in tissue and blood as well as on imaging in women at elevated risk for breast cancer. Twelve months after bariatric surgery, 50% of excess weight is generally expected. Eligible women at elevated risk for breast cancer who are already planning to undergo bariatric surgery will be consented to undergo imaging (MRI and mammogram), breast tissue biopsy, and fasting blood draw prior to bariatric surgery, approximately 14 days after bariatric surgery, and approximately 1 year after bariatric surgery.

In parallel we will also be assessing 40 normal breast tissue specimens as well as blood samples from the Komen Tissue Bank (elevated risk but normal BMI) to establish a normal BMI, elevated risk control group for our study. The KTB samples will be matched for general risk of breast cancer (>20%), age, race and menopausal status.

DETAILED DESCRIPTION:
Primary Objectives

1. The effect of bariatric surgery on Background Parenchymal Enhancement (BPE) on breast MRI through comparative analysis of images of women pre- and 1 year post-bariatric surgery.
2. The effect of bariatric surgery on breast density as seen on standard four view mammograms by qualitative BIRADS category through comparative analysis of images of women pre- and 1 year post-bariatric surgery.

   Secondary Objectives
3. The impact of bariatric surgery on obesity associated immune markers in breast tissue by:

   * Comparing cellular immune infiltrate components [B cells (CD 20), cytotoxic T cells (CD8), helper T cells (CD4), dendritic cells (CD11c), leukocytes (CD45), and monocytes/macrophages (CD68)] in breast tissue lobules of obese women pre-, 14 days post, and 1 year post bariatric surgery, and comparing these to normal breast tissue of lean women from the KTB
   * Comparing the presence of crown like structures (CLS) in breast tissue of obese women at pre-, 14 day post-, and 1 year post - bariatric surgery, and comparing these also to normal breast tissue of lean women from the KTB.
4. The effect of bariatric surgery on aromatase expression in breast tissue of obese women pre-, 14 day post-, and 1 year post-bariatric surgery, as compared to levels in breast tissue of lean women from KTB.
5. The effects of bariatric surgery on other blood correlatives pre- and 14 day and 1 year post-bariatric surgery including: 1) PGE2, TNF alpha, IL1 beta, IL-8 and IL-10 in the inflammatory pathway; 2) adiponectin, leptin, insulin, IGF1, and IGFBP3 in the insulin pathway; and 3) estradiol, SHBG, E2, T and DHEAS in the hormonal pathway. These will also be compared to blood samples from lean women in the KTB.

ELIGIBILITY:
Inclusion Criteria

1. Patients must be post-menopausal, defined as one of the following:

   1. Age over 60
   2. Prior oophorectomy
   3. No menstrual periods in the past 12 months without a medical procedure such as hysterectomy or uterine ablation
   4. FSH at castrate levels (> 40IU/L). Patients who do not meet criteria a-c (such as those under age 60 with prior hysterectomy but ovaries remain in place) will need to have an FSH level to confirm menopausal status prior to enrollment.
2. Patients must have a BMI ≥ 30 as calculated by the formula:

   Weight in pounds / height squared x 703 = BMI

   A BMI of:
   1. 18.5-24.9 is considered normal;
   2. 25.0-29.9 is considered overweight;
   3. 30.0+ is regarded as obese.
3. Patients must be planning to undergo primary bariatric surgery (no revisions).
4. Patients must be willing to provide a core tissue biopsy at baseline and with repeat tissue collection after 2 weeks and 12 months post-bariatric surgery.
5. Patients must be aged 18-75 years at the time of informed consent.
6. Patients must be accessible for treatment, adverse event tracking and follow-up as determined by the treating physician.
7. Patient consent and authorization for the release of health information must be obtained according to local institutional guidelines.

Exclusion Criteria

1. History of any malignancy except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years. History of breast cancer is not allowed.
2. Concurrent or planned participation in randomized trials of weight loss or exercise interventions or trials targeting insulin, IGF-1 or their receptors. These interventions would interfere with the endpoints.
3. Weight greater than 500 lbs at the time of imaging.
4. Known allergy to gadolinium which is used for MRI contrast.
5. History of life threatening allergic reaction to local anesthesia (lidocaine, xylocaine).
6. For the purposes of invasive breast biopsies, women must not have received therapeutic anticoagulation in the 1 month prior to enrollment, and must have no medical reason why post-operative prophylactic anticoagulation could be held for 12 hours (i.e. atrial fibrillation, history of deep venous thrombosis).
7. Prior history of breast irradiation.
8. Use of chemopreventatives such as tamoxifen or raloxifene at any time prior to enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study examining changes in female breast tissue pre and post-bariatric surgery.
Study Population: 20 total patients will be enrolled to the high risk/BMI > 30 cohort. Post-menopausal women are defined as: (1) those ≥ 50 years of age who had not menstruated during the preceding 12 months or who had castrate follicle-stimulating hormone levels (>40IU/L), (2) those who had undergone a bilateral oophorectomy.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in breast density via MRI from baseline | 1 year post-bariatric surgery
  Categorical measures will be reported numerically: 1-increased, 2-decreased, 3-no change
Change in breast density via mammography from baseline | 1 year post-bariatric surgery
  Categorical measures will be reported numerically: 1-increased, 2-decreased, 3-no change

SECONDARY OUTCOMES:
Comparison of number of crown-like structures in obese breast tissue and normal breast tissue | 14 days post-bariatric surgery
  Numerical measures
Comparison of number of crown-like structures in obese breast tissue and normal breast tissue | 1 year post-bariatric surgery
  Numerical measures
Change in aromatase expression markers in obese tissue from baseline | 14 days post-bariatric surgery
  Numerical measures
Comparison of aromatase expression markers in normal weight breast tissue with obese breast tissue | 14 days post-bariatric surgery
  Numerical measures
Change in aromatase expression markers in obese tissue from baseline | 1 year post-bariatric surgery
  Numerical measures
Comparison of aromatase expression markers in normal weight breast tissue with obese breast tissue | 1 year post-bariatric surgery
  Numerical measures
Change in other correlative blood markers (inflammatory, insulin, hormonal) from baseline | 14 days post-bariatric surgery
  Numerical measures
Change in other correlative blood markers (inflammatory, insulin, hormonal) from baseline | 1 year post-bariatric surgery
  Numerical measures

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (3):
- United States (3):
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana